CLINICAL TRIAL: NCT03578237
Title: Cryoanalgesia to Prevent Acute and Chronic Pain Following Surgery
Brief Title: Cryoanalgesia to Prevent Acute and Chronic Pain Following Surgery: A Randomized, Double-Masked, Sham-Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Epimed International (Industry); Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Cryo Prevention PILOTs
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Mastectomy; Upper Limb Amputation Below Elbow; Upper Limb Amputation Above Elbow; Lower Limb Amputation Below Knee; Lower Limb Amputation Above Knee; Knee Arthropathy; Shoulder Arthroplasty; Rotator Cuff Repair; Video-Assisted Thoracoscopic Surgery (VATS); Skin Grafting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only the investigator/physician applying the cryoneurolysis will be aware of the treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (active cryoneurolysis) (Experimental): Receiving active cryoneurolysis
  Interventions: Device: Cryoneurolysis (active)
- Sham (Sham Comparator): Receiving sham cryoneurolysis procedure
  Interventions: Device: Sham cryoneurolysis procedure

INTERVENTIONS:
Device: Cryoneurolysis (active) — Mastectomy (subjects 1-18): Myoscience Iovera device: full cryo cycle. Mastectomy (subjects 19-end) and all other procedures: Epimed PainBlocker device: 3 cycles of 2-minute gas activation separated by 1-minute defrost periods with an active probe which results in a decrease in temperature
  Arms: Treatment (active cryoneurolysis)
Device: Sham cryoneurolysis procedure — Mastectomy (subjects 1-18): Myoscience Iovera device: simulated full cryo cycle without administering gas to the probe.
  Mastectomy (subjects 19-end) and all other procedures: 3 cycles of 2-minute gas activation separated by 1-minute defrost periods with a SHAM probe that does not deliver gas to the tip or result in a drop in temperature
  Other Names: Placebo treatment
  Arms: Sham

SUMMARY:
The ultimate objective of the proposed line of research is to determine if cryoanalgesia is an effective adjunctive treatment for pain in the period immediately following various painful surgical procedures; and, if this analgesic modality decreases the risk of persistent postoperative pain, or "chronic" pain. The objective of the proposed pilot study is to optimize the protocol and collect data to power subsequent, definitive clinical trials.

Specific Aim 1: To determine if, compared with current and customary analgesia, the addition of cryoanalgesia decreases the incidence and severity of post-surgical pain.

Hypothesis 1a (primary): The severity of surgically-related pain will be significantly decreased on postoperative day 2 with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

Hypothesis 1b: The incidence of chronic pain will be significantly decreased one year following surgery with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

Hypothesis 1c: The severity of chronic pain will be significantly decreased one year following surgery with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

Specific Aim 2: To determine if, compared with current and customary analgesia, the addition of cryoanalgesia improves postoperative functioning.

Hypothesis 2a: Following primary unilateral knee and shoulder arthroplasty as well as rotator cuff repair, joint range of motion will be significantly increased within the year following surgery with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

Hypothesis 2b: Following video-assisted thoracoscopic surgery, inspiratory spirometry will be improved within the month following surgery with the addition of cryoanalgesia as compared with patients receiving solely standard-of-care treatment.

DETAILED DESCRIPTION:
Subjects will be individuals undergoing unilateral or bilateral mastectomy; upper or lower limb amputation; primary, unilateral total knee or shoulder arthroplasty; primary, unilateral rotator cuff repair; video-assisted thoracoscopic surgery; and burn-related skin grafting of the lateral thigh. Those who consent to participate in this study will have standard preoperative peripheral nerve blocks administered and catheters inserted: paravertebral blocks or a fascial plane block (e.g., erector spinae plane block) for mastectomy, femoral/sciatic for lower limb amputation, and brachial plexus (or terminal nerves) for upper limb amputation; femoral or adductor canal for total knee arthroplasty; interscalene for shoulder arthroplasty or rotator cuff repair; thoracic epidural for video-assisted thoracoscopic surgery (VATS); and lateral femoral cutaneous nerve for skin grafting of the lateral thigh.

Treatment group assignment (randomization). Subjects with successfully-administered peripheral nerve blocks (defined by sensory changes in the appropriate nerve distribution) will be allocated to one of two possible treatments:

1. cryoneurolysis
2. sham cryoneurolysis (placebo control)

Randomization will be stratified by surgery type (e.g., mastectomy, upper limb amputation, and lower limb amputation). Computer-generated randomization lists will be used to create sealed, opaque randomization envelopes with the treatment group assignment enclosed in each envelope labeled with the randomization number.

The specific nerves targeted will depend on the surgical site: intercostal nervesblocks (4 levels depending on the specific surgical approach) for mastectomy; femoral/sciatic for lower limb amputation, and brachial plexus (or terminal nerves) for upper limb amputation; infrapatellar branch of the saphenous nerve for knee arthroplasty; suprascapular nerve for shoulder surgery; intercostal nerves for VATS procedures, and the lateral femoral cutaneous nerve for skin grafting of the lateral thigh. The cryoneurolysis sites will be cleansed with chlorhexidine gluconate and isopropyl alcohol. Using the optimal ultrasound transducer for the specific anatomic location and subject anatomy (linear vs curvilinear array), the target nerves will be identified in a transverse cross-sectional (short axis) view.

We initially used a hand-held cryoneurolysis machine (Iovera, Myoscience, Redwood City, CA; prior to merger with Pacira Pharmaceuticals). For subjects randomized to sham, we inserted the angiocatheters just through the skin and subsequently place the probe through the angiocatheter, but not deeper than immediately subcutaneous (lidocaine 2% will be administered, as needed, to anesthetize the angiocatheter track). We simulated a cryo treatment but did not actually deliver gas to the probe. Therefore, there was no temperature change. However, since all subjects had a paravertebral block in place, and intercostal cryoneurolysis approach was via the subjects' back outside of their line of vision, subjects were unable to sense much besides the pressure of the angiocatheter insertion and remained masked to treatment group. For subjects randomized to receive cryoneurolysis, the same procedure was used, only the angiocatheters inserted deeper towards the intercostal nerves, the probes situated adjacent to the intercostal nerves, and active gas passed through the probe resulting in cryoneurolysis of the target nerves.

When it became available, the hand-held device was replaced by a console cryoneurolysis device. Cryoneurolysis probes are available for a console neurolysis device (PainBlocker, Epimed, Farmers Branch, Texas) that either (1) pass nitrous oxide to the tip inducing freezing temperatures; or, (2) vent the nitrous oxide at the base of the probe so that no gas reaches the probe tip, resulting in no temperature change. Importantly, these probes are indistinguishable in appearance, and therefore treating physicians, subjects, and all clinical staff will be masked to treatment group assignment [only the treating physician/investigator performing the cryoneurolysis with be unmasked]. An angiocatheter/introducer may be inserted beneath the ultrasound transducer and directed until the probe tip is immediately adjacent to the target nerve (lidocaine 2% will be administered, as needed, to anesthetize the angiocatheter track). The angiocatheter needle will be removed, leaving the angiocatheter through which the appropriate Epimed probe will be inserted until it is adjacent to the target nerve. The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation (active or sham) separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis. For the sham probes, the nitrous oxide will be vented prior to reaching the probe shaft, resulting in a lack of perineural temperature change. The process will be repeated with the same treatment probe for any additional nerves (e.g., all nerves will receive either active cryoneurolysis or sham/placebo, and not a mix of the two possible treatments).

Statistical Analysis. The limb amputation, total knee and shoulder arthroplasty, rotator cuff repair, VATS, and skin grafting subjects will be included in pilot studies to help power a future clinical trials, so the investigators will enroll a convenience sample and not have a pre-determined primary endpoint or statistical plan. However, the end points of most interest will be average pain score on postoperative day 2 for shoulder arthroplasty and skin grafting subjects, range-of-motion at 6 weeks for the rotator cuff repairs, range-of-motion for knee arthroplasty, and FEV1 for the VATS procedures.

For the subjects having mastectomy, the investigators will power this study for an acute pain end point which will provide conclusive results for that end point; but, the data will also be used to help power a subsequent large, multicenter clinical trial for a chronic pain-related end point (which will require far more subjects than the investigators will enroll for the current study).

For the mastectomy subjects, sample size calculations are centered around the hypothesis that cryoneurolysis decreases the incidence and severity of post-mastectomy pain in the week following surgery. To this end, the primary outcome is the average NRS (as administered as part of the Brief Pain Inventory) queried on the afternoon of postoperative day 2. The difference in the distribution of NRS between groups will be assessed using the Mann-Whitney U test. The investigators approximate power using the two-sample t-test. Assuming a standard deviation of 2.25 NRS points, and minimum clinically meaningful difference of 2 NRS points, n=30 patients per group provide 86% power with two-sided alpha=5%.

The t-test approximation was confirmed by simulating integer valued NRS scores in the range 0 to 10. One group was simulated by rounding normally distributed data with mean 1.5 and standard deviation 2.5 (resulting in median of 2 and interquartile range 0 to 3); and the other with mean 3.5 and standard deviation 2.5 (resulting in median of 4 and interquartile range 1 to 5). Note these resulting summary statistics are consistent with Ilfeld et al (2014). When 10,000 trials were simulated under these assumptions, the Mann-Whitney U test provided 89.5% power, and Type I error was maintained at 4.85%.

Differences between groups in demographic variables and secondary endpoints will be assessed with the Mann-Whitney U test for continuous or ordinal data, and Fisher's Exact test for categorical data. Box-and-whisker plots will be used to visualize distributions by group.

R version 3.4.4 (R-project.org) was used for sample size calculations and simulations; and the most recent version of R will be used at the time of analysis.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients of at least 18 years of age
2. scheduled for a primary, unilateral total knee or shoulder arthroplasty, primary unilateral rotator cuff repair, VATS procedure, skin grafting of the lateral thigh, unilateral or bilateral mastectomy, or limb amputation distal to the femoral/humeral head and including at least one metatarsal/metacarpal bone
3. single-injection or continuous peripheral nerve blocks block or epidural infusion planned for perioperative analgesia
4. accepting of a cryoneurolysis procedure

Exclusion Criteria:

1. chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
2. pregnancy
3. incarceration
4. inability to communicate with the investigators
5. morbid obesity (body mass index > 40 kg/m2)
6. possessing any contraindication specific to cryoneurolysis such as a localized infection at the treatment site, cryoglobulinemia, cold urticaria and Reynaud's Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ilfeld, MD, MS, Principal Investigator — University California San Diego; John Finneran, MD, Study Director — University California San Diego; Matthew Swisher, MD, MS, Study Director — University California San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ACTIVE Cryoneurolysis: Receiving active cryoneurolysis
  Cryoneurolysis (active): Mastectomy (subjects 1-18): Myoscience Iovera device: full cryo cycle.
  Mastectomy (subjects 19-end) and all other procedures: Epimed PainBlocker device: 3 cycles of 2-minute gas activation separated by 1-minute defrost periods with an active probe which results in a decrease in temperature
- SHAM Cryoneurolysis: Receiving sham cryoneurolysis procedure
  Sham cryoneurolysis procedure: Mastectomy (subjects 1-18): Myoscience Iovera device: simulated full cryo cycle without administering gas to the probe.
  Mastectomy (subjects 19-end) and all other procedures: 3 cycles of 2-minute gas activation separated by 1-minute defrost periods with a SHAM probe that does not deliver gas to the tip or result in a drop in temperature
Period: Postoperative Days 0-21
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Started | 51 | 48
Completed | 51 | 48
Not Completed | 0 | 0
Period: Postoperative Day 0 - Month 12
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Started | 51 | 48
Completed | 37 | 32
Not Completed | 14 | 16
Not completed — Timepoints past 21 days were only for amputee and mastectomy subjects and not others | 14 | 16

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Active Cryoneurolysis): Receiving active cryoneurolysis
  Cryoneurolysis (active): Mastectomy (subjects 1-18): Myoscience Iovera device: full cryo cycle.
  Mastectomy (subjects 19-end) and all other procedures: Epimed PainBlocker device: 3 cycles of 2-minute gas activation separated by 1-minute defrost periods with an active probe which results in a decrease in temperature
- Sham: Receiving sham cryoneurolysis procedure
  Sham cryoneurolysis procedure: Mastectomy (subjects 1-18): Myoscience Iovera device: simulated full cryo cycle without administering gas to the probe.
  Mastectomy (subjects 19-end) and all other procedures: 3 cycles of 2-minute gas activation separated by 1-minute defrost periods with a SHAM probe that does not deliver gas to the tip or result in a drop in temperature
- Total: Total of all reporting groups
Arm/Group | Treatment (Active Cryoneurolysis) | Sham | Total
Number analyzed (Participants) | 51 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (15) | 52 (16) | 51.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 31 | 71
  Male | 11 | 17 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kilograms] | 70.6 (13.7) | 68.8 (14.8) | 69.6 (14.2)
Height [Mean (Standard Deviation); unit: centimeters] | 165.1 (8.0) | 165.7 (7.6) | 165.4 (7.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (4.6) | 25.0 (4.5) | 25.4 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Average Pain (Mastectomy Subjects Only)
Description: Measured with the 0-10 numeric rating scale as part of the Brief Pain Inventory, with 0 equivalent to no pain and 10 equivalent to the worst imaginable pain
Time Frame: afternoon of postoperative day 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 51 | 48
score on a scale | 0.0 [0 to 1.4] | 3.0 [2.0 to 5.0]

2. Secondary Outcome: Analgesic Consumption
Description: Analgesic consumption for previous 24 hours
Time Frame: Postoperative days 1, 2, 3, 4, 7, 14, 21, as well as months 1, 3, 6, and 12
Measure: Mean (Standard Deviation); unit: tablets of oxycodone (5 mg tablets)
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 51 | 48
tablets of oxycodone (5 mg tablets)
  Postoperative Day 1 | 1.2 (2.3) | 3.3 (4.5)
  Postoperative Day 2 | 1.0 (1.6) | 4.1 (3.8)
  Postoperative Day 3 | .8 (1.9) | 3.2 (3.7)
  Postoperative Day 4 | 0.7 (1.5) | 2.7 (3.5)
  Postoperative Day 7 | 0.5 (1.2) | 1.5 (2.2)
  Postoperative Day 14 | 0.2 (0.6) | 0.5 (1.3)
  Postoperative Day 21 | 0.1 (0.5) | 0.3 (0.8)
  Postoperative Month 1 | 0 (0) | 0 (0)
  Postoperative Month 3 | 0 (0) | 0 (0)
  Postoperative Month 6 | 0 (0) | 0 (0)
  Postoperative Month 12 | 0 (0) | 0 (0)

3. Secondary Outcome: Brief Pain Inventory (Interference Subscale)
Description: The Brief Pain Inventory short form (interference scale) is designed to assess pain's impact on physical and emotional functioning. It has established reliability and validity, with minimal inter-rater discordance, and is recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus statement. The interference domaine is comprised of 7 questions involving the degree of pain's interference on physical and emotional functioning using a 0-10 Likert scale (0 = none; 10 = complete). The scale is thus 0-70 with higher scores equivalent to more interference due to pain>
Time Frame: Months 1, 3, 6, and 12
Population: mastectomy and amputee participants only (other participants did not have outcome measures collected for these time points)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 37 | 32
units on a scale
  Month 1 | 0 (0) | 4.1 (9.2)
  Month 3 | 0 (0) | 0.6 (2.9)
  Month 6 | 0 (0) | 1.1 (2.3)
  Month 12 | 0 (0) | 0.3 (0.9)

4. Secondary Outcome: Worst Pain Measured on the 11 Point Numeric Rating Scale
Description: The subjects' perception of their worst level pain in the previous 24 hours measured with the 0-10 numeric rating scale as part of the Brief Pain Inventory, with 0 equivalent to no pain and 10 equivalent to the worst imaginable pain
Time Frame: Postoperative days 1, 2, 3, 4, 7, 14, and 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 51 | 48
score on a scale
  Postoperative Day 1 | 3.7 (2.5) | 5.5 (2.4)
  Postoperative Day 2 | 3.3 (2.9) | 5.6 (2.7)
  Postoperative Day 3 | 2.8 (2.7) | 5.1 (2.8)
  Postoperative Day 4 | 2.4 (2.6) | 4.3 (2.7)
  Postoperative Day 7 | 2.4 (2.4) | 3.7 (2.4)
  Postoperative Day 14 | 1.6 (2.4) | 3.1 (2.3)
  Postoperative Day 21 | 1.4 (2.6) | 3.0 (2.5)

5. Secondary Outcome: Average Pain Measured on the 11 Point Numeric Rating Scale
Description: The subjects' perception of their average level pain in the previous 24 hours measured with the 0-10 numeric rating scale as part of the Brief Pain Inventory, with 0 equivalent to no pain and 10 equivalent to the worst imaginable pain
Time Frame: Postoperative days 1, 2, 3, 4, 7, 14, and 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 51 | 48
score on a scale
  Postoperative day 1 | 1.5 (1.8) | 3.2 (2.1)
  Postoperative day 2 | 1.5 (2.0) | 3.3 (1.9)
  Postoperative day 3 | 1.2 (2.1) | 2.8 (1.9)
  Postoperative day 4 | 1.2 (2) | 2.4 (1.9)
  Postoperative day 7 | 0.8 (1.3) | 2 (1.9)
  Postoperative day 14 | 0.9 (1.9) | 1.6 (1.5)
  Postoperative day 21 | .7 (1.5) | 1.6 (1.8)

6. Secondary Outcome: Difficultly Sleeping Due to Pain
Description: Difficulty sleeping due to pain (binary answer: yes or no; not based on a scale or instrument). The numbers presented in the results are the number of participants in each treatment group answering YES, they DID have difficulty sleeping due to pain
Time Frame: Postoperative days 1, 2, 3, 4, 7, 14, and 21
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 51 | 48
Participants
  Postoperative day 1 | 5 | 11
  Postoperative day 2 | 6 | 11
  Postoperative day 3 | 6 | 13
  Postoperative day 4 | 3 | 10
  Postoperative day 7 | 4 | 11
  Postoperative day 14 | 4 | 7
  Postoperative day 21 | 4 | 7

7. Secondary Outcome: Number of Awakenings
Description: Number of awakenings from sleep due to pain (simply the number of times of awakenings--not based on a scale or instrument)
Time Frame: Postoperative days 1, 2, 3, 4, 7, 14, and 21
Measure: Mean (Standard Deviation); unit: Awakenings
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 51 | 48
Awakenings
  Postoperative day 1 | 0.1 (0.6) | .8 (1.4)
  Postoperative day 2 | .3 (1) | .5 (1)
  Postoperative day 3 | .4 (1.2) | .9 (1.6)
  Postoperative day 4 | .3 (.9) | .5 (.8)
  Postoperative day 7 | .1 (.4) | .5 (1)
  Postoperative day 14 | .3 (1) | .3 (.6)
  Postoperative day 21 | .2 (.9) | .4 (.9)

8. Secondary Outcome: Nausea
Description: Nausea measured on a 0-10 scale with 0=no nausea and 10=vomiting; thus higher on the scale is worse
Time Frame: Postoperative days 1, 2, 3, 4, 7, 14, and 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 51 | 48
units on a scale
  Postoperative day 1 | .5 (1.5) | .6 (2.1)
  Postoperative day 2 | .1 (.5) | .3 (.9)
  Postoperative day 3 | 0 (0) | 0.3 (1.1)
  Postoperative day 4 | .2 (1.1) | .1 (.9)
  Postoperative day 7 | .1 (.3) | .3 (1.7)
  Postoperative day 14 | 0 (0) | 0 (0)
  Postoperative day 21 | 0 (0) | 0 (0)

9. Secondary Outcome: Phantom Pain Occurences [Mastectomy & Amputation]
Description: How many times in the previous 3 days subject experienced phantom pain (the number of times experienced--not based on a scale or instrument)
Time Frame: Postoperative months 1, 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Occurrences
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 37 | 32
Occurrences
  Month 1 | 0 (0) | 0.5 (1.8)
  Month 3 | 0 (0) | 9.8 (2.5)
  Month 6 | 0 (0) | 4.0 (1.9)
  Month 12 | 0 (0) | 0.4 (1.2)

10. Secondary Outcome: Phantom Pain Duration [Mastectomy & Amputation]
Description: The average duration of phantom pain occurrences in the previous 3 days
Time Frame: Postoperative months 1, 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 37 | 32
hours
  Month 1 | 0 (0) | 0.1 (0.2)
  Month 3 | 0 (0) | 0 (0.2)
  Month 6 | 0 (0) | 5.1 (20.1)
  Month 12 | 0 (0) | 0 (0.2)

11. Secondary Outcome: Phantom Sensation Occurrences [Mastectomy & Amputation]
Description: How many times in the previous 3 days subject experienced phantom sensations (the number of times experienced--not based on a scale or instrument). This outcome differs from "phantom pain occurrences" in that for this outcome no pain is necessary; rather, participants feel the missing body part is actually there, when it is not--yet it is not a painful sensation.
Time Frame: Postoperative months 1, 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: incidences
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 37 | 32
incidences
  Month 1 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 1.2 (3.1)
  Month 6 | 0 (0) | 0.5 (1.7)
  Month 12 | 0 (0) | 10.3 (26.7)

12. Secondary Outcome: Phantom Sensation Duration [Mastectomy & Amputation]
Description: The average duration of phantom sensation occurrences in the previous 3 days. This outcome differs from "phantom pain duration" in that for this outcome no pain is necessary; rather, participants feel the missing body part is actually there, when it is not--yet it is not a painful sensation.
Time Frame: Postoperative months 1, 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 37 | 32
hours
  Month 1 | 0 (0) | 0 (0)
  Month 3 | 0 (0) | 0.1 (0.3)
  Month 6 | 0 (0) | 1.7 (8.9)
  Month 12 | 0 (0) | 7.8 (26.8)

13. Secondary Outcome: Residual Limb or Wound Pain Occurences
Description: How many times in the previous 3 days subject experienced residual limb or wound pain (the number of times experienced--not based on a scale or instrument)
Time Frame: Postoperative months 1, 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Occurrences
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 37 | 32
Occurrences
  Month 1 | 0.9 (1.6) | 20 (37.1)
  Month 3 | 0 (0) | 4.4 (18.4)
  Month 6 | 0.1 (0.4) | 5.3 (18.4)
  Month 12 | 0.1 (0.4) | 1.1 (3.4)

14. Secondary Outcome: Residual Limb or Wound Pain Duration
Description: The average duration of residual limb or wound pain occurrences in the previous 3 days
Time Frame: Postoperative months 1, 3, 6, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
Number analyzed (Participants) | 37 | 32
hours
  Month 1 | 0.1 (0.3) | 17.6 (37.8)
  Month 3 | 0 (0) | 3.5 (18.4)
  Month 6 | 0 (0.2) | 5.3 (20.1)
  Month 12 | 0 (0) | 0 (0.2)

ADVERSE EVENTS:
Time Frame: Mastectomy participants: 1 year Amputation participants: 1 year Burn participants: 21 days Total knee arthroplasty participants: 21 days
Arm/Group | ACTIVE Cryoneurolysis | SHAM Cryoneurolysis
All-Cause Mortality (participants affected / at risk) | 0/51 | 2/48
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 0/51 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03578237/Prot_SAP_000.pdf